CLINICAL TRIAL: NCT00535587
Title: Maximizing Exercise Effectiveness in Fibromyalgia
Brief Title: Testing Mestinon and Exercise in Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Kim Dupree Jones PhD, Associate Professor, Oregon Health & Science University, School of Nursing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R01NR008150-04 (NIH); R01NR008150 (NIH)
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Exercise; Mestinon
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Exercise; Pyridostigmine Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental)
  Interventions: Behavioral: Exercise; Drug: pyridostigmine
- 2 (Experimental)
  Interventions: Drug: pyridostigmine; Drug: Placibo
- 3 (Experimental)
  Interventions: Behavioral: Exercise; Behavioral: Attention Control
- 4 (Experimental)
  Interventions: Drug: Placibo; Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Exercise
  Arms: 1; 3
Drug: pyridostigmine
  Other Names: Mestinon
  Arms: 1; 2
Drug: Placibo
  Arms: 2; 4
Behavioral: Attention Control
  Arms: 3; 4

SUMMARY:
The purpose of this trial was to test the combined and independent effects of 6 months of exercise and Mestinon in people with fibromyalgia. Specifically, we wanted to determine if Mestinon helped people with fibromyalgia have an easier time exercising and if their symptoms improved by the end of the trial.

DETAILED DESCRIPTION:
Earlier, we demonstrated that people with fibromyalgia fail to make adequate growth hormone when they exercise intensively. We also demonstrated that a single dose of Mestinon helped people make normal levels of growth hormone when they exercised in our laboratory. We wanted to know if 6 months of exercise with concurrent Mestinon therapy would make growth hormone (and related markers) normal and improve fibromyalgia symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Have Fibromyalgia

Exclusion Criteria:

* Subjects will be excluded if they have a history of rheumatic disease or other disorder that may compromise ability to safely complete study protocol, be pregnant, nursing, or currently involved in unresolved litigation.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2002-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edit Serfozo, MPH, Study Director — Oregon Health and Science University; Kim Dupree Jones, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mestinon & Exercise | Mestinon and Attention Control | Placebo Pill and Exercise | Placebo Pill and Attention Control
Started | 53 | 53 | 47 | 54
Completed | 43 | 42 | 39 | 41
Not Completed | 10 | 11 | 8 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mestinon & Exercise | Mestinon and Attention Control | Placebo Pill and Exercise | Placebo Pill and Attention Control | Total
Number analyzed (Participants) | 53 | 53 | 47 | 54 | 207
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 53 | 47 | 54 | 207
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49 (9) | 49 (8) | 50 (7) | 49 (8) | 49 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 49 | 45 | 54 | 201
  Male | 0 | 4 | 2 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 53 | 53 | 47 | 54 | 207

OUTCOME MEASURES:

1. Primary Outcome: Levels of Growth Hormone Post Exercise
Description: Serum growth hormone at peak V02/treadmill
Time Frame: 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Mestinon/Exercise | Placebo Pill/Attention Control
Number analyzed (Participants) | 43 | 41
ng/ml | 4.95 (3.07) | 1.41 (2.94)
Statistical Analysis 1: Comparison: Mestinon/Exercise vs Placebo Pill/Attention Control; Test type: Superiority or Other; p < 0.02, ANCOVA; Median Difference (Final Values) = .05, Standard Deviation 2.94

2. Secondary Outcome: Improvement of Fibromyalgia Symptoms
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Mestinon & Exercise | Mestinon and Attention Control | Placebo Pill and Exercise | Placebo Pill and Attention Control
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/36 | 0/39 | 0/41
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/39 | 0/41

LIMITATIONS AND CAVEATS:
6 discontinued due to medical reasons unrelated to the study 4 were unwilling to complete

1 relocated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes